CLINICAL TRIAL: NCT01764932
Title: Determining the Accuracy of Thoracic Epidural Continuous Catheter Insertion With Confirmatory Fluoroscopic Imaging
Brief Title: Accuracy of the Thoracic Epidural Catheter Insertion Confirmed by Fluoroscopic Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chicago Anesthesia Pain Specialists (Other)
Responsible Party: Principal Investigator, Kenneth D Candido, Chairman of the Anesthesia Department, Advocate Illinois Masonic Medical Center, Chicago Anesthesia Pain Specialists
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Advocate-IRB-5242
Record Dates: First submitted 2013-01-02; First posted 2013-01-10 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Patients Undergoing Thoracic Surgery; Patients Undergoing Upper Abdominal Surgery

ARMS (1):
- Thoracic epidural catheter insertion (Other): Fluoroscopic imaging. For patients undergoing thoracic epidural analgesia (TEA) with catheter placement for pain associated with thoracic or upper abdominal surgery
  Interventions: Procedure: Fluoroscopic imaging

INTERVENTIONS:
Procedure: Fluoroscopic imaging — Contrast media (5 mL) will be injected through the catheter and fluoroscopic images will be obtained and saved in the lateral and antero-posterior projections.

SUMMARY:
In patients scheduled for thoracic surgery or upper abdominal surgery, investigators will determine the accuracy of the epidural catheter placement by using fluoroscopic imaging.

Previous studies have drawn contradictory conclusions based the potential flaw assumption of 100% success rate for correct epidural catheter placement in the thoracic region.

DETAILED DESCRIPTION:
Thoracic epidural analgesia (TEA) is a key tool in management of pain after thoracic or upper abdominal surgery. TEA optimizes pain relief while minimizing the use of systemic opioids, thus reducing the duration of postoperative ileus. TEA also attenuates surgical stress response and allows for early mobilization. Despite all the touted benefits of TEA, much controversy limits its use for post surgical pain due to fear of exceedingly rare, if not entirely theoretical complication of epidural hematoma.

Beneficial effects of TEA require that catheter placement and infusate be targeted at the thoracic segments innervating injured skin, muscle, and bone from which pain input originates. The purpose of this study is to determine the accuracy of thoracic epidural continuous catheter insertion by using fluoroscopic imaging.

ELIGIBILITY:
Inclusion Criteria:

* 18- 80 years old patients
* Patients undergoing thoracic surgery
* Patients undergoing upper abdominal surgery

Exclusion Criteria:

* Severe Aortic Valve stenosis
* Active Neurologic Disease
* Allergy to lidocaine or bupivacaine
* Allergy to iodine-based contrast
* Cutaneous Disorders at epidural insertion site
* Preoperative impaired coagulation status
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-12; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Presumed intervertebral level of epidural catheter | During procedure
  At the time of thoracic epidural catheter insertion

SECONDARY OUTCOMES:
Radiologic confirmation of epidural catheter placement | Post procedure within one week.
  Radiology department will assess within one week after the procedure the images, to confirm the epidural catheter placement.
Change in Numeric Rating Pain Score from baseline | 1, 24 and 48 hrs
  1, 24, and 48 hrs after the end of the surgery.

OTHER OUTCOMES:
Patient satisfaction | Post procedure at 48 hours
  Patient satisfaction 48 hrs after the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Candido, M.D., Principal Investigator — Chicago Anesthesia Pain Specialists
Locations (1):
- Advocate Illinois Masonic Medical Center, Chicago, Illinois, United States